CLINICAL TRIAL: NCT03217786
Title: Early Post Transplant Cardiac Allograft Vasculopathy
Acronym: ECAV
Status: Active, not recruiting | Type: Observational
Sponsor: Ottawa Heart Institute Research Corporation (Other)
Collaborators: Toronto General Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 0868
Record Dates: First submitted 2017-07-11; First posted 2017-07-14 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-04

CONDITIONS: Cardiac Allograft Vasculopathy
Keywords: Macrovascular Disease; Microvascular Coronary Artery Disease; Cardiac Transplant Rejection; Transplant; Failure, Heart; Intravascular ultrasound (IVUS); Optical Coherence Tomography; Index of Microcirculatory Resistance; Fractional Flow Reserve; Coronary Flow Reserve; Positron Emission Tomography; Endomyocardial Biopsies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Specimens will be assessed for potential CAV biomarkers.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Heart transplantation is an effective life-saving treatment for patients with end-stage heart disease. After a transplant, the new heart may develop narrowing in the arteries, causing heart failure, heart attacks and abnormal heart rhythms. This condition is known as cardiac allograft vasculopathy (CAV). The disease is very common, affecting almost a third of heart transplant patients by 5 years after transplant. CAV is a serious problem that causes the new heart to fail and is one of the main causes of death after transplant. Early detection of CAV is important as treatment options are poor once the disease is established. Currently, available techniques to evaluate CAV are limited by poor ability to detect disease early. The current tests usually focus on the large heart arteries and do not examine the smaller arteries that are also affected.

DETAILED DESCRIPTION:
The objective of this study is to determine whether early abnormalities of the heart arteries after heart transplantation can predict the development of CAV. We will use a combination of sophisticated imaging tools to examine in detail the early changes that occur in the arteries of a new heart. Heart transplant patients from the University of Ottawa Heart Institute and Toronto General Hospital will undergo a series of tests at 3 and 12 months after transplant. Statistical analyses will determine whether results from the above tests at 3 months predict the development of early CAV at 12 months after a heart transplant.

ELIGIBILITY:
Inclusion Criteria:

1. Heart transplant <3 months.
2. Age ≥18 years.
3. Able and willing to provide informed consent.

Exclusion Criteria:

1. Contraindications to dipyridamole.
2. Contraindications to aminophylline.
3. Contraindications to nitroglycerin.
4. Contraindications to iodinated contrast.
5. Acute allograft rejection ≤1 month.
6. Uncontrolled heart failure or myocardial infarction ≤7 days.
7. Estimated glomerular filtration rate ≤30 mL/min.
8. Combined solid organ transplantation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This prospective longitudinal study will involve 2 Canadian adult heart transplant programs: University of Ottawa Heart Institute (UOHI, Ottawa) and University Health Network-Toronto General Hospital (UHN-TGH, Toronto).
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2018-02-12 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
CAV on invasive coronary studies | 3 months and 1-year post-transplant.
  Changes in coronary intima on IVUS and OCT and invasive coronary flow

SECONDARY OUTCOMES:
EMBx | 3 months post-transplant
  Microvascular disease
PET | 3 months post-transplant
  Myocardial blood flow quantification
Biomarkers | 3 months post-transplant
  Serum biomarker panel

CONTACTS AND LOCATIONS:
Overall Officials: Sharon Chih, MD, PhD, Principal Investigator — Ottawa Heart Institute Research Corporation
Locations (1):
- University of Ottawa Heart Institute, Ottawa, Ontario, Canada

REFERENCES:
- [Derived] Chih S, Tavoosi A, Nair V, Chong AY, Dzavik V, Aleksova N, So DY, deKemp RA, Amara I, Wells GA, Bernick J, Overgaard CB, Celiker-Guler E, Mielniczuk LM, Stadnick E, McGuinty C, Ross HJ, Beanlands RSB. Cardiac PET Myocardial Blood Flow Quantification Assessment of Early Cardiac Allograft Vasculopathy. JACC Cardiovasc Imaging. 2024 Jun;17(6):642-655. doi: 10.1016/j.jcmg.2023.10.003. Epub 2023 Nov 22. PMID 37999656
- [Derived] Chih S, Chong AY, Dzavik V, So DY, Aleksova N, Wells GA, Bernick J, Overgaard CB, Stadnick E, Mielniczuk LM, Beanlands RSB, Ross HJ. Fibrotic Plaque and Microvascular Dysfunction Predict Early Cardiac Allograft Vasculopathy Progression After Heart Transplantation: The Early Post Transplant Cardiac Allograft Vasculopathy Study. Circ Heart Fail. 2023 Jun;16(6):e010173. doi: 10.1161/CIRCHEARTFAILURE.122.010173. Epub 2023 May 11. PMID 37165901